CLINICAL TRIAL: NCT03931564
Title: SIGHT Study: Cost-effectiveness of InnFocus Microshunt (IMS) Implantation Versus Standard Trabeculectomy (TE)
Brief Title: SIGHT Study: Cost-effectiveness of InnFocus Microshunt Implantation vs. Trabeculectomy.
Acronym: SIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL68964.068.19
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-10

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Glaucoma, Open-Angle; Trabeculectomy; Intraocular Pressure; Minimally invasive glaucoma surgery; InnFocus Microshunt; PRESERFLO Microshunt
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESERFLO Microshunt (formerly InnFocus Microshunt (IMS)) (Active Comparator): The intervention group will undergo PRESERFLO (formerly InnFocus) Microshunt implantation (IMS).
  Interventions: Procedure: PRESERFLO Microshunt implantation
- Trabeculectomy (Active Comparator): The usual care/control group will undergo a standard trabeculectomy.
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: PRESERFLO Microshunt implantation — The intervention consists of the microshunt implantation augmented with mitomycin C application.
  Other Names: InnFocus Microshunt implantation
  Arms: PRESERFLO Microshunt (formerly InnFocus Microshunt (IMS))
Procedure: Trabeculectomy — The usual care / control group will undergo a standard fornix based trabeculectomy augmented with mitomycin C application.
  Arms: Trabeculectomy

SUMMARY:
The standard surgical treatment for glaucoma is trabeculectomy. The PRESERFLO™ (formerly InnFocus) Microshunt (IMS) is a new, minimally invasive drainage device which has been suggested to result in similar IOP lowering, but with faster visual recovery and less complications and postoperative interventions. The objective of this study is to aid in deciding on the use of the IMS in glaucoma surgery by assessing its efficacy and cost-effectiveness in patients with primary open angle glaucoma (POAG) compared to the standard trabeculectomy (TE).

DETAILED DESCRIPTION:
During the last decade, minimally invasive glaucoma surgery (MIGS) procedures have been introduced to the market. MIGS procedures or devices, often small stents or tubes that can be placed into the eye, are potentially safer than standard trabeculectomy (TE). The surgery is faster and easier to perform. Patient recovery is faster with fewer postoperative visits, suggesting less impact on vision and quality of life. However, MIGS devices are more expensive compared to standard surgery and it is unclear if the higher costs can be compensated with their better safety profile and faster patient recovery (reduced productivity losses).

To establish guidelines for the use of MIGS, the Netherlands Glaucoma Group has recognized the need for a formal investigation of their cost-effectiveness as compared to TE, prior to their implementation on a large scale for regular care. Therefore, a societal cost-effectiveness analysis of MIGS procedures will be undertaken to further elucidate their position in the glaucoma treatment algorithm in the Netherlands.

The objective of this study is to aid in deciding on the use of the IMS in glaucoma surgery by assessing its efficacy and cost-effectiveness in patients with primary open angle glaucoma compared to trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Caucasian patients aged between 18 and 80 years old with uncontrolled primary open angle glaucoma on (maximum tolerated) medical therapy and/or progression of visual field loss, an IOP ≥18 and ≤40 mmHg, and an indication for primary glaucoma surgery (trabeculectomy) are suitable for inclusion.

Exclusion Criteria:

1. Patient unwilling or unable to give informed consent, unwilling to accept randomization or inability to complete follow-up (e.g. hospital visits) or comply with study procedures
2. Secondary glaucoma (e.g. pigment dispersion syndrome, pseudo exfoliation syn-drome, iris neovascularization, rubeosis iridis, trauma, epithelial or fibrous down growth, iridocorneal endothelial syndrome, etcetera).
3. Previous incisional surgery of the subject eye. Previous uncomplicated clear corneal cataract surgery is allowed >6 months prior to the surgery.
4. Poor vision in either the study or fellow eye. Poor vision is defined as a corrected vis-ual acuity <0.6 and/or a visual field loss within the central 10 degrees (with exception of a superior altitudinal defect).
5. Any ocular comorbidities that could affect the visual field. (e.g. diabetic retinopathy, proliferative retinopathy, aphakia, degenerative visual disorder not associated with glaucoma)
6. Chronic or recurrent uveitis.
7. Need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery.
8. Anatomical factors that increase the risk of complicated surgery (due to previous trauma, anatomical abnormalities, anterior synechiae or previous cyclodestructive procedure).
9. Conditions that increase the risk of endophthalmitis.

   * Current ocular, adnexal or periocular infections (e.g., untreated blepharitis)
   * Immune compromised patients including the use of topical or systemic steroids for an indication other than the surgery within 3 months of the procedure (this would not include the use of inhaled or dermatologic steroids), chemotherapy within 6 months of the procedure.
   * Iodine allergy
   * Unwilling to discontinue contact lens after surgery
10. Contraindication or allergy to mitomycin C.
11. Any contraindication to tube placement (e.g. shallow anterior chamber, insufficient endothelial cell density).
12. Use of oral hypotensive glaucoma medications for treatment of the fellow eye.
13. Prior ocular laser treatment within 3 months of the surgery, increasing the risk of in-flammation in the eye.
14. Corneal thickness <450um or >620microns.
15. Conditions associated with elevated episcleral venous pressure such as active thyroid orbitopathy.
16. Among patients in whom both eyes are eligible only the first eye is undergoing surgical treatment is enrolled in the study.
17. Participation in another clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 12 months postoperatively
  The intraocular pressure is measured using a Goldmann applanation tonometer

SECONDARY OUTCOMES:
Visual acuity | baseline, 1 week, 4 weeks, 3, 6, 9 and 12 months postoperatively
  Measured with ETDRS letter charts
Glaucoma medical therapy | at baseline and 1 day, 1 week, 4 weeks, 3, 6, 9 and 12 months postoperatively
  number of glaucoma drugs (active substances)
Failure rate | 3, 6, 9 and 12 months postoperatively
  Failure is defined as an IOP >21 mmHg and ≤ 5 mmHg or less than 20% reduction relative to baseline IOP at two consecutive follow-up visits after 3 months. Reoperation will also be defined as failure.
Complications | Intraoperatively and up to 12 months after the surgery.
  The incidence of intraoperative and postoperative complications.
Reinterventions | Measured up to 12 months after the surgery.
  The number of reinterventions after the surgery.
Visual field progression | measured twice at baseline and twice after 12 months of follow-up.
  The progression seen on the visual field.
Mean endothelial cell loss | measured at baseline and after 12 months of follow-up.
  The endothelial cell density will be measured using specular microscopy photography.
Patient- reported outcome measures (PROMs): NEI-VFQ-25 | measured at baseline, 4 weeks, 3, 6, and 12 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by National Eye Institute Visual Function Questionnaire (NEI VFQ-25).
Patient- reported outcome measures (PROMs): GQL-15 | measured at baseline, 4 weeks, 3, 6, and 12 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by Glaucoma Quality of Life-15 (GQL-15).
Patient- reported outcome measures (PROMs): EuroQol's EQ-5D-5L | measured at baseline, 4 weeks, 3, 6, and 12 months postoperatively
  Health-related quality of life as measured by EuroQol's EQ-5D-5L questionnaire.
Patient- reported outcome measures (PROMs): HUI3 | measured at baseline, 4 weeks, 3, 6, and 12 months postoperatively
  Health-related quality of life as measured by HUI3 (Health Utility Index Mark 3) questionnaire.
Quality Adjusted Life Years (QALYs) | Baseline until 12 months postoperatively
  Calculated based on generic health-related quality of life, using the EQ-5D-5L and HUI-3 questionnaires
Costs per patient | Baseline until 12 months postoperatively
  Cost per patient, including valuation of resource use by using the Dutch guidelines for cost-analyses or cost prices provided by the medical center.
Incremental cost-effectiveness ratios (ICERs): QALY | Baseline until 12 months postoperatively
  Evaluation of cost-effectiveness by using calculated costs per quality-adjusted life years (QALYs)
Incremental cost-effectiveness ratios (ICERs): NEI VFQ-25 | Baseline until 12 months postoperatively
  Calculated costs per clinically improved patient on the NEI VFQ-25 questionnaire
Incremental cost-effectiveness ratios (ICERs): GQL-15 | Baseline until 12 months postoperatively
  Calculated costs per clinically improved patient on the GQL-15 questionnaire
Incremental cost-effectiveness ratios (ICERs): IOP | Baseline until 12 months postoperatively
  Calculated costs per patient with clinically lowered IOP
Budget impact | Baseline until 12 months postoperatively
  Reported as a difference in costs. Different scenario's will be compared to investigate the impact of various levels of implementation (e.g. 25%, 50%, 75% of eligible patients).

CONTACTS AND LOCATIONS:
Overall Officials: Henny Beckers, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+ (MUMC+), Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scheres LMJ, van den Biggelaar FJHM, Winkens B, Kujovic-Aleksov S, Muskens RPHM, de Waard PWT, de Crom RMPC, Ernest PJG, Pijl BJ, Ramdas WD, van Rijn LJ, Tan A, Dirksen CD, Beckers HJM. Effectiveness and cost-effectiveness of MicroShunt implantation versus standard trabeculectomy for open-angle glaucoma (a SIGHT study): study protocol of a multicentre randomised controlled trial. BMC Ophthalmol. 2023 Jan 31;23(1):43. doi: 10.1186/s12886-022-02734-y. PMID 36721130